CLINICAL TRIAL: NCT05435170
Title: A Phase I, Randomized, Open-label, Single Dose, 2 Period, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of Linerixibat Tablets in Healthy Adult Participants
Brief Title: Food Effect Study of Linerixibat Tablets in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 214656
Expanded Access: NCT05448170 (Available)
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Pruritus
Keywords: Pharmacokinetic; Pharmacodynamic; Food effect; Ileal bile acid transporter (IBAT) inhibitor; Linerixibat
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the 2 sequences. In sequence AB, participants will receive linerixibat under fed state (Treatment A) in Period 1, then linerixibat under fasted state (Treatment B) in Period 2. In Sequence BA, the 2 treatments will be reversed. The washout period will be of at least 7 days.
Masking Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence AB (Experimental): Participants will receive linerixibat in fed state (Treatment A) in period 1 followed by linerixibat in fasted state (Treatment B) in period 2. The washout period will be of at least 7 days.
  Interventions: Drug: linerixibat
- Treatment sequence BA (Experimental): Participants will receive linerixibat in fasted state (Treatment B) in period 1 followed by linerixibat in fed state (Treatment A) in period 2. The washout period will be of at least 7 days.
  Interventions: Drug: linerixibat

INTERVENTIONS:
Drug: linerixibat — linerixibat will be administered per the treatment sequence

SUMMARY:
This study will evaluate the effect of food on the Pharmacokinetic (PK) and Pharmacodynamic (PD) parameters of linerixibat administered in fed and fasted states in heathy adult participants

ELIGIBILITY:
Inclusion criteria:

* Overtly healthy male or female participants 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants' age greater than (>) 50 years old, must have had at least 3 weeks elapsed after the completion of an approved primary SARS-CoV-2 vaccination course.
* Body weight >50 kg and body mass index (BMI) within the range 18.5 - 32 kilogram per meter square (kg/m2) (inclusive).
* Female Participants:

  * A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:
  * Is a woman of non-childbearing potential (WONCBP). OR
  * Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year).
* Capable of giving signed informed consent.

Exclusion Criteria:

* History of cholecystectomy.
* Current symptomatic cholelithiasis or inflammatory gall bladder disease.
* Significant history of or current disorders capable of significantly altering the absorption, metabolism, or elimination of drugs.
* Current clinically significant diarrhea.
* History of gastrointestinal surgery with ileal resection or ileal bypass at any time.
* Any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Administration of any other Ileal Bile Acid Transport (IBAT) inhibitor (including linerixibat) in the 3 months prior to screening.
* Past or intended use of over the counter or prescription medication, including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inhibitor) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless approved by the Investigator in conjunction with GSK Medical Monitor.
* Current enrollment in a clinical trial or recent participation in a clinical trial and has received an investigational product within the following time period prior to study drug administration: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months before the first dose in the current study.
* Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5x upper limit of normal (ULN).
* Bilirubin >1.5x ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody test or hepatitis C Ribonucleic acid (RNA) test at screening or within 3 months prior to first dose of study intervention.
* Positive human immunodeficiency virus (HIV) antibody test
* Fridericia's QT correction formula (QTcF) >450 msec on ECG performed at screening.
* Regular use of known drugs of abuse or history of drug abuse or dependence within 6 months of the study.
* Regular alcohol consumption within 6 months prior to signing the informed consent.
* Regular use of tobacco- or nicotine-containing products in the 3 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Plasma linerixibat area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration [AUC(0-t)] | Up to 36 hours post dose
Maximum observed plasma concentration (Cmax) of linerixibat | Up to 36 hours post dose

SECONDARY OUTCOMES:
Plasma linerixibat area under the concentration-time curve from time zero (pre-dose) to infinite time [AUC (0-∞)] | Up to 36 hours post dose
Plasma linerixibat area under the concentration-time curve from time zero (pre-dose) to 24 hour [AUC (0-24)] | Up to 24 hours post dose
Time of occurrence of Cmax (Tmax) of linerixibat | Up to 36 hours post dose
Delay in achieving Tmax (Tlag) of linerixibat | Up to 36 hours post dose
Apparent terminal phase half-life (t1/2) of linerixibat | Up to 36 hours post dose
Apparent clearance (CL/F) of linerixibat | Up to 36 hours post dose
Apparent terminal phase volume of distribution (Vz/F) of linerixibat | Up to 36 hours post dose
Serum C4 area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration [AUC(0-t)] | Up to 36 hours post dose
Serum C4 area under the concentration-time curve from time zero (pre-dose) to 24 hour [AUC (0-24)] | Up to 24 hours post dose
Incidence of adverse events (AEs) and of serious adverse events (SAEs) | Up to day 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinincal Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.